CLINICAL TRIAL: NCT07225777
Title: Sex Differences in Neurobehavioral Response to Acute THC in Adults With Cannabis Use Disorder
Brief Title: Sex Differences in Neurobehavioral Response to THC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin Martin, Research Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00148223; K12DA031794 (NIH)
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use Disorder
Keywords: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Males (Other)
  Interventions: Drug: Dronabinol; Drug: Placebo
- Females (Other)
  Interventions: Drug: Dronabinol; Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Oral dronabinol capsules (40 mg)
  Other Names: Marinol
Drug: Placebo — Matched placebo capsules

SUMMARY:
This study investigates sex differences in reward processing following acute THC administration in adults with cannabis use disorder (CUD). Using multimodal neuroimaging (MRS and fMRI), the study will assess glutamate levels in the nucleus accumbens and striatal BOLD response to monetary reward anticipation. Participants will complete two counterbalanced dosing sessions (oral THC 40 mg vs. placebo).

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45
* DSM-5 criteria for CUD
* Cannabis use ≥4 days/week
* THC-positive urine
* BMI 18-30
* Regular menstrual cycle (females)
* Willingness to use non-hormonal birth control (females)

Exclusion Criteria:

* Lifetime psychotic or bipolar disorder
* Recent drug use other than cannabis
* Current psychotropic medication
* Treatment-seeking for SUD
* Current psychiatric disorder (except mild alcohol, nicotine, or caffeine use disorder)
* Pregnancy/nursing
* MRI contraindications

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Nucleus accumbens glutamate | 2 hours post-dose
  Concentrations of nucleus accumbens glutamate measured via proton magnetic resonance spectroscopy
Striatal reward anticipation | 3 hours post-dose
  Blood oxygen-level-dependent (BOLD) signaling in the striatum (caudate, putamen, nucleus accumbens) measured using functional magnetic resonance imaging (fMRI) during a monetary reward task

SECONDARY OUTCOMES:
Drug Effects Questionnaire (DEQ) - Like Drug Effect | 0-7 hours
  Visual Analog Scale rating of subjective drug liking included in the Drug Effects Questionnaire. Score ranges from 0 (not at all) to 100 (extremely) using a 100mm line anchored with none/extreme designation.
Drug Effects Questionnaire (DEQ) - Want More | 0-7 hours
  Visual Analog Scale rating of subjective desire for more of the same drug included in the Drug Effects Questionnaire. Score ranges from 0 (not at all) to 100 (extremely) using a 100mm line anchored with none/extreme designation.
Drug Effects Questionnaire (DEQ) - High | 0-7 hours
  Visual Analog Scale rating of subjective "high" included in the Drug Effects Questionnaire. Score ranges from 0 (not at all) to 100 (extremely) using a 100mm line anchored with none/extreme designation.
Nucleus accumbens GABA | 2 hours post-dose
  Concentrations of nucleus accumbens GABA measured via proton magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Erin Martin, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States